CLINICAL TRIAL: NCT04301544
Title: Filipino Multicomponent Intervention to Maintain Cognitive Performance in High Risk Population (FINOMAIN): Integration of Complementary Non-Pharmacological Approach With Standard Medical Care for Elderly With Cognitive Impairment
Brief Title: Filipino Multicomponent Intervention to Maintain Cognitive Performance in High Risk Population (FINOMAIN)
Acronym: FINOMAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Luke's Medical Center, Philippines (Other)
Collaborators: Nanyang Technological University (Other); Icahn School of Medicine at Mount Sinai (Other); University of Copenhagen (Other)
Responsible Party: Principal Investigator, Jacqueline C. Dominguez, MD, Head, Memory Center, St. Luke's Medical Center, Philippines
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CT-18146; PITAHC-IDxxx (Other: PITAHC)
Record Dates: First submitted 2020-02-13; First posted 2020-03-10 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild Cognitive Impairment (MCI); Multicomponent intervention; Dance; Vascular risk factors
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INDAK & Standardized Vascular Care Group (Experimental): The experimental arm will receive training on the ballroom dance modules called INDAK (Improving Neurocognition through Dance and Kinesthetics), nutrition counseling and vascular risk management
  Interventions: Behavioral: INDAK (Improving Neurocognition through Dance and Kinesthetics); Behavioral: Nutrition Counseling; Behavioral: Standardized Vascular Care
- Standardized Vascular Care Group (Active Comparator): The control group will receive nutrition counseling and vascular risk management
  Interventions: Behavioral: Nutrition Counseling; Behavioral: Standardized Vascular Care

INTERVENTIONS:
Behavioral: INDAK (Improving Neurocognition through Dance and Kinesthetics) — INDAK (Improving Neurocognition through DAnce and Kinesthetics) is a structured modular dance consisting of 8 types of ballroom dances (Reggae, Cha-cha, Samba, Merengue, Bachata, Swing, Tango and Salsa) with increasing complexity. The intervention group will receive dance intervention from a dance teacher two times a week, one hour each time, for 12 months. Each 60-minute session has 3 parts: 10 minutes warm-up/ stretching, 40 minutes dance proper and 10 minutes cool down. This dance intervention will last for 12 months.
  Other Names: INDAK
  Arms: INDAK & Standardized Vascular Care Group
Behavioral: Nutrition Counseling — The dietary advice will follow Filipino Nutrition Research Institute (FNRI) recommendation called Pinggang Pinoy or Filipino Plate, which is a picture of a nine-inch plate with foods proportionally distributed among the food groups to provide approximately 1,200 to 1,500 calories per day. It is advised that half of the plate is composed of green leafy vegetables and one serving of fruit per meal. For fruits, 4 to 6 servings are encouraged per day. In general, affordable nutritious food is recommended: high consumption of local fruits and vegetables, brown/purple rice instead of white rice, coconut oil and other vegetable oils, and fish. Participants will be asked to use structured 3-day meal diary for diet monitoring. Individual counseling sessions depending on identified vascular risks based on FNRI recommendations will also be conducted. This is followed-up by study nutritionists every 3-month of intervention period.
Behavioral: Standardized Vascular Care — The management advice for hypertension, diabetes, and dyslipidemia will be based on Filipino standard clinical practice guidelines. This is followed-up by study physicians every 3-month of intervention period

SUMMARY:
FINOMAIN is a community-based, cluster randomized controlled trial (cRCT) of dance intervention INDAK and standardized vascular care. The study aims to develop and assess the effectiveness of a cost-effective and culturally - fit intervention for Filipino older adults at high risk for developing dementia.

The first objective of the study is to evaluate the efficacy of dance intervention INDAK on cognitive function as assessed by the Alzheimer's Disease Assessment Scale - Cognitive (ADAS-Cog), Mnemonic Similarity Task (MST), and Executive Function Composite (EFC) among older adults with mild cognitive impairment (MCI). To increase the sensitivity of primary outcome for various composites of cognition, aside from ADAS-Cog that assesses core cognitive deficits of dementia, investigators will develop an executive function composite that will combine measures of executive control using performance outcomes on tests including Trail Making Test (TMT), Digit Symbol Substitution Test (DSST), Verbal Fluency Test (VFT), and Number Cancellation Task (NCT). Executive function composite scores have been used to track aging populations at risk for dementia and are shown to be sensitive in capturing cerebrovascular benefits and used as instruments in studies with similar non-pharmacological intervention (i.e. aerobic exercise, dance). Additionally, the investigators will add MST which is a measure for episodic memory, memory representations and pattern discrimination which are all cognitive domains highly correlated with hippocampal function.

The second objective of the study is to determine the effect of dance on neuroplasticity as measured by brain volumetry and functional connectivity demonstrated through Magnetic Resonance Imaging (MRI) and change in other behavioral and functional outcomes of participants with MCI.

DETAILED DESCRIPTION:
FINOMAIN is a single-blind (assessor blinded), community-based, cluster randomized controlled trial (cRCT) of a multi-component intervention with two arms. The intervention arm will receive 12 months (1 hour, 2 times per week) of training on the ballroom dance modules called INDAK (Improving Neurocognition through Dance and Kinesthetics), nutrition counseling, and vascular risks management. The control group will receive the same nutrition counseling and vascular risk management except for dance (INDAK).

Study population: In this pilot trial of FINOMAIN, the study aims to enroll at least 72 (20% of total sample size of 328) community-dwelling Filipino older adult participants aged 60 years and above with mild cognitive impairment (MCI) based on Petersen criteria and documented by cognitive symptoms and cognitive performance on the standardized cognitive test (ADAS-Cog) which is ≥ 1.5 standard deviation (SD) below Filipino norms for ADAS-Cog and has a Clinical Dementia Rating (CDR) of 0.5. Participants should not fulfill DSM-V criteria for major neurocognitive disorders. The absence of dementia is further confirmed when there is no functional impairment based on the Lawton's Instrumental Activities of Daily Living (IADL) scale and no significant neuropsychiatric symptoms as detected by the Neuropsychiatric Inventory - Questionnaire (NPI-Q). Exclusion to study are major sensory impairment (i.e. hearing and visual impairment) that limit testing, dance participation and a pre-existing illness that in the judgment of the study physician precludes engagement in moderate physical activity such as INDAK.

The study duration will be 24 months, but the study intervention will last for 12 months. The intervention arm will receive 12 months (1 hour, 2 times per week) of training on the dance modules called INDAK, nutrition counseling and vascular risks management. The control group will receive the same nutrition counseling and vascular risk management except dance (INDAK).

The intervention team consists of research nurses, nutritionists, physicians and dance teachers. The dance intervention INDAK is a structured modular dance consisting of 8 types of ballroom dances with increasing complexity. The INDAK intervention will be done two times a week, one hour each time, for 12 months. The nurse will use a logbook to register the frequency and duration of participation for each participant. From our previous experience, adverse events were infrequently limited to musculoskeletal pains in the first two weeks of study. However, to ensure safety, a trained nurse will always be present at each dance session and liaise with local hospitals in case of unexpected events such as fall, dizziness, or general exhaustion occur. The nurse records the vital signs of all participants before and after the dance.

The nutrition counseling is based on "Pinggang Pinoy" or Filipino plate recommendation of the Filipino Nutrition Research Institute (FNRI) and standardized vascular care for hypertension, diabetes, and dyslipidemia based on Filipino standard guidelines. The nurses will monitor the participants every month and use a logbook to record their compliance and advise participants on a continuing basis. The community physicians and nurses will meet with the participants at 3, 6, and 9 months to monitor their cardiovascular and metabolic conditions and revise their management plan if necessary. If the nurses detect an urgent problem during the monthly monitoring, nurses must alert participants to see the community physicians on an ad-hoc basis. The participants will also be provided with a diary to log their implementation of risk management plans and issues that need to be discussed with the nurses and physicians.

Follow-up visits will be conducted by the assessment team (i.e. neurologists, psychologists and nurses) on the 6th and 12th month of the intervention. To ensure blinding, participants are asked not to discuss any intervention with anyone. At each meeting, the same clinical data as from the baseline assessments and laboratory tests will be collected as mentioned above. Neuroimaging will be done 12 months from baseline. After all data are collected and encoded, data cleaning, processing, and analysis will be done. The following are the methods for data acquisition, processing, and analysis:

MRI acquisition, processing, and analysis: Participants will be scanned in a 3T MRI scanner (Philips Achieva) using an 8-channel head coil. The ADNI-3 (http://adni.loni.usc.edu/adni-3/) recommended imaging protocols will be used to allow data to be comparable with the ADNI centers and good potential for data sharing on open access platforms. For resting-state fMRI, participants will be asked to keep their eyes open and fixate on a cross (10 minutes). The fMRI task: Participants will undergo 2 runs (6 -7 minutes each) of the visual working memory task. Each cycle consists of 1 block of high-load and 1 block of low-load that had 2 trials each. Each block is interleaved by a 1.6 seconds interval and block duration of 20 seconds. There will be 10 cycles in each run adding up to a total of 20 high-load and 20 low-load trials. Each run lasts 400 seconds.

Voxel-Based Morphometry (VBM8) will be applied for overall brain volumetric analysis with the high-resolution MPRAGE T1-weighted image acquisition. FMRIB Software Library (FSL) and Tract Based Spatial Statistics (TBSS) will be applied for diffusion MRI to understand changes in structural connectivity. The high-resolution MPRAGE scan will also be applied for automated hippocampal volumetric studies using NeuroQuant. Coronal axial thin T2-weighted and FLAIR will be used for detecting subcortical and deep white mater hyperintensities (WMH). The fMRI data will be pre-processed and analyzed using the Statistical Parametric Mapping (SPM12) software package. All structural and functional images will be re-oriented before the EPI data is pre-processed using the conventional procedure in three phases.

Statistical Analysis (Neurocognitive and behavioral measures): The primary outcome which is the change from baseline (ADAS-Cog, MST, and EFC which a composite of Verbal Fluency Test (VFT), Number Cancellation Task (NCT), Digit Symbol Substitution Task (DSST) and Trail Making Test (TMT) and the secondary outcomes (neuroimaging: MRI, GDS, EQVAS BBS) will be analyzed in the intent-to-treat population as well as in the per-protocol population (complete at least 80% of INDAK modules and participate in at least 30 minutes of dance each time). The study will employ univariate, bivariate, and multivariate statistics. For univariate, descriptive statistics (mean/SD; frequencies/percentages) will be used to summarize socio-demographic and other baseline characteristics. The bivariate analyses that examine underlying relationships between the outcomes and other clinical characteristics are the following: t-test for continuous variables and Chi-square test (or Fisher Exact Test when 20 of the cells have the expected count less than five) for categorical variables to compare baseline data and outcome measures at baseline between the intervention and control groups. For multivariate analyses, the study would estimate the effect from baseline to follow-up at 12 months between randomization groups. Since the participants will be measured 3 times (baseline, 6 months, 12 months), the study will be using the repeated measures analysis of covariance (RM ANCOVA) to test the significance between group means but controlling for possible confounders. To analyze for the secondary outcomes, the power will be calculated retrospectively to see if the sample size is big enough to prove statistical significance. Assuming that enough power is yielded, repeated measures ANCOVA will also be used.

The end of study analysis will be done for three months and the final report will be prepared for three months to answer the aims of the study on how multicomponent intervention significantly maintains or improve cognition of older adults with MCI as measured by primary outcomes and how the intervention affects neural plasticity and functional connectivity as measured by MRI after 12 months of the study period.

ELIGIBILITY:
Inclusion criteria:

* Aged ≥ 60 years old
* Mild cognitive impairment (MCI) based on Petersen criteria
* Standardized cognitive test ≥1.5 standard deviation (SD) below norms
* Do not fulfill DSM-V criteria for major cognitive disorders
* Clinical Dementia Rating (CDR) of 0.5

Exclusion criteria:

* Significant functional impairment based on Lawton's IADL
* Significant neuropsychiatric impairment based on NPI-Q
* Significant hearing and visual impairment that limit testing and dance participation
* Pre-existing illness that in the judgment of the study physician precludes engagement in moderate physical activity

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2019-05-28 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Alzheimer's Disease Assessment Scale - Cognitive Score | At 6th month and 12th month of intervention
  To measure the cognitive function in Alzheimer's disease (AD), hence its popularity for use in cognitive testing of the effects of AD treatment in clinical trials. It consists of 11 tasks measuring the core cognitive deficits of AD, such as disturbances of memory, language, praxis, attention, visuospatial function and other cognitive abilities. ADAS-Cog was validated for use in the Filipino elderly with age and education stratified norms. Score ranges from 0 to 70 points, with lower scores indicating better cognitive functions.
Change from baseline in Mnemonic Similarity Task score | At 6th month and 12th month of intervention
  This task place strong demands on pattern separation, memory representation and measures cognitive domains highly correlated with hippocampal function. Pre-MST use set 1, self-paced timing, consisting two phases: encoding and test part. The encoding phase presents 128 colored photographs of objects on computer screen (2 secs duration; ≥ 0.5 secs inter-stimulus-interval/ISI) to be classified by participants as either indoor (key "V") or outdoor (key "N"). The test phase consists of 192 items (64 repeated items, 64 lure items and 64 foil items; presented 2 secs, ≥ 0.5 secs ISI), in which participants engaged in a modified recognition task identifying each item as Old (key "V"), Similar (key "B") or New (key "N"). Percentage accuracy is calculated, with higher percentage indicating better functions.
Change from baseline in Executive Function Composite score | At 6th month and 12th month of intervention
  To evaluate fluency, attention, visual scanning, processing and psychomotor speed.

SECONDARY OUTCOMES:
Change from baseline in Magnetic Resonance Imaging (MRI) | At 12th month of intervention
  To evaluate structural and functional connectivity of the brain
Change from baseline in Brief Geriatric Depression Scale (GDS) score | At 6th month and 12th month of intervention
  To evaluate depressive symptoms. GDS score ranges from 0 to 15, with lower scores indicating less depressive symptoms.
Change from baseline in Change in EuroQoL - Visual Analog Scale (EQVAS) rating | At 6th month and 12th month of intervention
  EQVAS is used as self-rated scale. The scores range from 0 to 100, with higher rates indicating better perception of health related quality of life.
Change from baseline in Change in Berg Balance Scale (BBS) score | At 6th month and 12th month of intervention
  To measure for balance. BBS consist of 14 tasks where participants are asked to sit, stand, move or reach using different stance like using standing on one leg, eyes close, turning and reaching forward or backward. The score ranges from 0 to 56, with higher scores indicating better functions.

OTHER OUTCOMES:
Compliance | At 6th and 12th month of intervention
  Defined as 80% attendance to dance exercise (INDAK) with completion of full 60-minute dance sessions, as well as attendance to vascular risk factor intensive monitoring and management visits done by team of nurse, physician and nutritionist.

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline C Dominguez, MD, Principal Investigator — St. Luke's Medical Center
Locations (1):
- Institute for Neurosciences, St. Luke's Medical Center, Quezon City, National Capital Region, Philippines